CLINICAL TRIAL: NCT00915018
Title: A Randomized, Open-Label, Two-Arm Study Of Neratinib Plus Paclitaxel Versus Trastuzumab Plus Paclitaxel As First-Line Treatment For ErbB-2-Positive Locally Recurrent Or Metastatic Breast Cancer
Brief Title: Study Evaluating Neratinib Plus Paclitaxel VS Trastuzumab Plus Paclitaxel In ErbB-2 Positive Advanced Breast Cancer
Acronym: NEFERTT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3144A2-3005 / B1891005
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer
Keywords: ErbB-2 positive advanced breast cancer; HKI-272; Neratinib; Nerlynx; HER2; PB-272; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — neratinib; Trastuzumab; Paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- neratinib plus paclitaxel (Experimental)
  Interventions: Drug: Neratinib; Drug: Paclitaxel
- trastuzumab plus paclitaxel (Active Comparator)
  Interventions: Drug: Trastuzumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Neratinib — Neratinib - 240 mg orally daily, administered once daily. Treatment will be administered until documented disease progression, symptomatic deterioration, unacceptable toxicity, death or withdrawal of consent.
  Arms: neratinib plus paclitaxel
Drug: Trastuzumab — Trastuzumab - 4 mg/kg IV initial loading dose followed by subsequent once weekly doses of 2mg/kg IV. Treatment will be administered until documented disease progression, symptomatic deterioration, unacceptable toxicity, death or withdrawal of consent.
  Other Names: Herceptin; Herclon
  Arms: trastuzumab plus paclitaxel
Drug: Paclitaxel — Paclitaxel - 80 mg/m² IV administered on days 1, 8, and 15 of a 28-day cycle. Treatment will be administered until documented disease progression, symptomatic deterioration, unacceptable toxicity, death or withdrawal of consent.
  Other Names: Taxol; Abraxane; Onxol; Nov-onxol

SUMMARY:
This study is investigating the effects of an experimental drug (neratinib) in combination with paclitaxel versus trastuzumab in combination with paclitaxel for the treatment of women who have not received previous treatment for erbB-2-positive locally recurrent or metastatic breast cancer. The study will compare the effectiveness of each regimen in shrinking tumors and extending the lives of women with erbB-2 (HER2) positive breast cancer. The study will also compare the safety of the two regimens and as well as the quality of life of subjects receiving either regimen.

ELIGIBILITY:
Inclusion Criteria:

* ErbB-2 positive locally recurrent or metastatic breast cancer
* Eastern Cooperative Oncology Group (ECOG) 0-2
* Measurable disease
* Availability of tumor tissue for HER2 status confirmation

Exclusion Criteria:

* Prior systemic anti-cancer therapy other than endocrine therapy for locally recurrent or metastatic disease
* Prior erbB-2 inhibitor other than trastuzumab or lapatinib in the neoadjuvant or adjuvant setting
* Progression/recurrence within 12 months after completion of adjuvant or neoadjuvant therapy
* History of heart disease
* History of gastrointestinal disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 479 (Actual)
Dates: Start 2009-08-21 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2018-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Puma, Study Director — Biotechnology
Locations (195):
- United States (36):
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - Redwood Regional Medical Group, Santa Rosa, California
  - Cancer Center of Central Connecticut, Plainville, Connecticut
  - Palm Beach Institute of Hematology and Oncology, Boynton Beach, Florida
  - North Broward Medical Center Cancer Center, Deerfield Beach, Florida
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Mid Florida Cancer Centers, Orange City, Florida
  - Florida Cancer Research Institute, Plantation, Florida
  - Hematology Oncology Associates of Treasure Coast, Port Saint Lucie, Florida
  - Phoebe Cancer Center, Albany, Georgia
  - Dublin Hematology and Oncology Care, Dublin, Georgia
  - Clintell, Skokie, Illinois
  - Presence Hematology and Oncology, Skokie, Illinois
  - Springfield Clinic, Springfield, Illinois
  - CHRISTUS St. Frances Cabrini Hospital, Alexandria, Louisiana
  - Hematology Oncology Services, Metairie, Louisiana
  - Park Nicollet Institute, Saint Louis Park, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - St. John's Medical Research Institute, Springfield, Missouri
  - Washington University School of Medicine Siteman Cancer Center, St Louis, Missouri
  - The Valley Hospital, Luckow Pavilion Office of Oncology Clinical Trials, Paramus, New Jersey
  - Gaston Hematology and Oncology Associates, Gastonia, North Carolina
  - Summa Health System Hospitals, Akron, Ohio
  - Warren Cancer Research Foundation, Tulsa, Oklahoma
  - Samaritan Hematology and Oncology Consultants, Corvallis, Oregon
  - Pawtucket Memorial Hospital, Pawtucket, Rhode Island
  - Medical University of South Carolina Hollings Cancer Center, Charleston, South Carolina
  - Santee Hematology Oncology, Sumter, South Carolina
  - Tenessee Cancer Specialists, Knoxville, Tennessee
  - Family Cancer Care, Memphis, Tennessee
  - Texas Oncology, Bedford, Texas
  - El Paso Cancer Treatment Center, El Paso, Texas
  - Texas Oncology-Allison Cancer Center, Midland, Texas
  - Southlake Oncology, Southlake, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Charleston Area Medical Center, Health, Education, and Research Institute, Charleston, West Virginia
- Australia (2):
  - The Queen Elizabeth Hospital, North Adelaide, South Australia
  - Royal Melbourne Hospital, Parkville, Victoria
- Belarus (4):
  - N.N. Aleksandrov National Cancer Center of Belarus, Lyasny, Minsk Oblast
  - Institution of Healthcare Grodno Regional Clinical Hospital, Grodno
  - Institution Gomel Regional Clinical Oncology Dispensary, Homyel
  - Healthcare Institution Vitebsk Regional Clinical Oncology Dispensary, Vitebsk
- Institut Jules Bordet, Brussels, Belgium
- Bulgaria (3):
  - District Dispensary for Oncology Diseases Internal Unit- Plovdiv EOOD, Plovdiv
  - District Dispensary for Oncology Diseases Internal Unit- Sofia EOOD, Sofia
  - Specialised Hospital of ActiveTreatment in Oncology, Clinic of Chemotherapy, Sofia
- Canada (2):
  - Hopital Charles, LeMoyne Le Centre Intégré de Cancérologie de la Montérégie, Greenfield Park, Quebec
  - Centre Hospitalier Régional de Trois-Rivières, Trois-Rivières, Quebec
- China (9):
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangdong
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing
  - Peking Union Medical College Hospital of Chinese Academy of Medical Sciences, Beijing
  - The Hospital Affiliated Academy Military Medical Science, Chinese People's Liberation Army, Beijing
  - Chinese People's Liberation Army General Hospital, Beijing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Cancer Hospital, Tianjin
- Croatia (2):
  - Clinical Hospital Osijek, Department of Radiotherapy and Oncology, Osijek
  - University Hospital For Tumors, Zagreb
- Rigshospitalet, Copenhagen, Onkologisk Klinik, Copenhagen, Denmark
- France (11):
  - Hôpital Henri-Mondor, Créteil
  - Centre Leon Berard Departement de Cancerologie Medicale, Lyon
  - Centre Val d'Aurelle, Montpellier
  - Hopital Hotel Dieu, Service d'Oncologie Medicale, Bat B2, 5ieme, Paris
  - Hopital La Pitie-Salpetriere, Paris
  - Groupe Hospitalier Paris Saint Joseph, Oncologie medicale, Paris
  - Service d'Oncologie et de Radiotherapie, Polyclinique Francheville, Périgueux
  - Clinique Armoricaine de Radiologie, Saint-Brieuc
  - Centre de Radiothérapie, Clinique Sainte Anne, Service d'Oncologie Libérale, Strasbourg
  - CHU Strasbourg Departement Oncologie & Hematologie Hopital Civil, Strasbourg
  - CHU Bretonneau, Centre Henry Kaplan, Tours
- Sozialstiftung Bamberg Klinik fuer Haematologie und internistische Onkologie, Bamberg, Germany
- Hong Kong (3):
  - Pamela Youde Nethersole Eastern Hospital, Chai Wan
  - Queen Mary Hospital, Hong Kong
  - UNIMED Medical Institute, Comprehensive Centre for Breast Diseases, Wan Chai
- Hungary (7):
  - Semmelweis Egyetem Radiologiai és Onkoterapias Klinika, Budapest
  - Fovarosi Onkormanyzat Szent Imre Korhaz Klinikai Onkologiai Profil, Budapest
  - Orszagos Onkologiai Intezet "B" Belgyogyaszati osztaly, Budapest
  - Kaposi Mor Oktato Korhoz Onkologiai Centrum, Kaposvár
  - Bacs-Kiskun Megyei Onkormanyzat Korhaza Onkoradiologiai Kozpont, Kecskemét
  - Borsod-Abaúj-Zemplén Megyei Kórház és Egyetemi Oktató Kórház, Miskolc
  - Szegedi Tudomanyegyetem Onkoterapias Klinika, Szeged
- India (10):
  - Jawaharlal Nehru Cancer Hospital, Bhopal, Madhya Pradesh
  - Tata Memorial Centre, Mumbai, Maharashtra
  - Central India Cancer Research Institute, Nagpur, Maharashtra
  - Curie Manavata Cancer Centre, Nashik, Maharashtra
  - Shatabdi Super Speciality Hospital, Nashilk, Maharashtra
  - Deenanath Mangeshkar Hospital and Research Centre, Pune, Maharashtra
  - Institute Rotary Cancer Hospital, AIIMS, New Delhi, National Capital Territory of Delhi
  - Searoc Cancer Center, Jaipur, Rajasthan
  - Meenakshi Mission Hospital and Research Centre, Madurai, Tamil Nadu
  - B P Poddar and Medical Research Ltd., Kolkata, West Bengal
- Israel (3):
  - Kaplan Medical Center, Rehovot
  - Sourasky Medical Center, Tel Aviv
  - Assaf Harofeh Medical Center, Ẕerifin
- Italy (5):
  - Policlinico di Modena Oncologia ed Ematologia, Modena
  - Fondazione Salvatore Maugeri, Pavia
  - Policlinico Universitario Campus Bio-Medico, Roma
  - Ospedale San Pietro Fatebenefratelli, Roma
  - Ospedale San Giovanni Battista-Molinette, Torino
- Japan (33):
  - Hyogo Cancer Center, Hyōgo, Akashi-shi
  - National Hospital Organization Beppu Medical Center, Ōita, Beppu-shi
  - Tokyo Metropolitan Cancer and Infectious Disease Center, Komagome Hospital, Tokyo, Bunkyo-ku
  - Chiba Cancer Center, Chiba, Chiba-shi
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka-shi
  - National Hospital Organization Mito Medical Center, Ibaraki, Higashiibaraki-gun
  - Hiroshima University Hospital, Hiroshima, Hiroshima-shi
  - Hakuaikai Medical Corporation Sagara Hospital, Kagoshima, Kagoshima-city
  - National Cancer Center Hospital East, Chiba, Kashiwa-shi
  - Saitama Cancer Center, Saitama, Kitaadachi-gun
  - Kumamoto Municipal Hospital, Kumamoto, Kumamoto-city
  - Kurume Daiichi Social Insurance Hospital, Fukuoka, Kurume-Shi
  - National Hospital Organization Shikoku Cancer Center, Ehime, Matsuyama-city
  - Iwate Medical University Hospital, Numakunai, Morioka-shi
  - Aichi Cancer Center, Aichi, Nagoya-shi
  - National Hospital Organization Nagoya Medical Center, Aichi, Nagoya
  - Niigata Cancer Center Hospital, Niigata, Niigata-shi
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka, Osaka-shi
  - National Hospital Organization Osaka National Hospital, Osaka, Osaka-shi
  - National Hospital Organization Hokkaido Cancer Center, Hokkaido, Sapporo-shi
  - Tohoku University Hospital, Miyagi, Sendai-city
  - Tenri Hospital, Nara, Tenri-shi
  - Kanagawa Cancer Center, Kanagawa, Yokohama-City
  - Hiroshima City Hospital, Hiroshima
  - National Hospital Organization Kure Medical Center and Chugoku Cancer Center, Hiroshima
  - Kobe City Medical Center General Hospital, Hyōgo
  - Shinko Hospital, Hyōgo
  - Kumamoto University Hospital, Kumamoto
  - Tazuke Kofukai Medical Research Institute Kitano Hospital, Osaka
  - Osaka University Hospital, Osaka
  - Jichi Medical University Hospital, Tochigi
  - Toranomon Hospital, Tokyo
  - National Hospital Organization Tokyo Medical Center, Tokyo
- Latvia (3):
  - Piejuras Hospital, Liepajas Oncological Clinic, Liepāja
  - Pauls Stradiņš Clinical University Hospital, Riga
  - Riga Eastern University Hospital, Riga
- Lithuania (2):
  - Hospital of Lithuanian University of Health sciences, Kaunas
  - Nacionalinis Vezio Institutas, Vilniaus Universiteto Onkologijos Institutas, Vilnius
- University Malaya Medical Centre, Kuala Lumpur, Malaysia
- Sir Anthony Oncology Center, Floriana, Malta
- Poland (5):
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Szpital Wojewodzki Oddzial, Jelenia Góra, Lower Silesian Voivodeship
  - Magodent, Warsaw, Masovian Voivodeship
  - Opolskie Centrum Onkologii, Opole, Opole Voivodeship
  - Zakład Opieki Zdrowotnej MSW z Warmińsko, Mazurskim Centrum Onkologii, Olsztyn, Warmian-Masurian Voivodeship
  - Białostockie Centrum Onkologii, Bialystok
- Hospital da Luz Servico de Oncologia Medica, Lisbon, Portugal
- Romania (3):
  - Institutul Oncologic Prof. Dr. Ion Chiricuţă, Cluj-Napoca, Cluj
  - SC Oncolab S.R.L., Craiova, Dolj
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
- Serbia (2):
  - Institute of Oncology and Radiology of Serbia, Belgrade
  - Clinical centre Nis Clinic of Oncology, Niš
- Singapore (2):
  - National University Hospital, National Cancer Institute, Singapore
  - National Cancer Centre Singapore, Singapore
- South Africa (7):
  - GVI Oncology, Port Elizabeth, Eastern Cape
  - The Medical Oncology Centre of Rosebank, Johannesburg, Gauteng
  - University of Witwatersrand Oncology, Donald Gordon Medical Centre, Johannesburg, Gauteng
  - Sandton Oncology Centre, Johannesburg, Gauteng
  - Eastleigh Breast Care Centre, Pretoria, Gauteng
  - Westridge Medical Centre, Durban, KwaZulu-Natal
  - GVI Oncology, Kraaifontein, Western Cape
- South Korea (5):
  - National Cancer Center, Center for Breast Cancer, Goyang-si, Gyeonggi-do
  - Samsung Medical Center, Seoul, Korea
  - Asan Medical Center, Seoul, Korea
  - Korea University Guro Hospital, Seoul, Korea
  - Yonsei University Health System Severance Hospital, Seoul, Seoul/Korea
- Spain (12):
  - Hospital Son Llàtzer, Palma, Balearic Islands
  - Hospital Universitari Arnau de Vilanova, Lleida, Catalonia
  - Complejo Hospitalario Universitario Santiago de Compostela, Santiago de Compostela, Galicia
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Puerta De Hierro, Majadahonda, Madrid
  - Hospital Universitario Infanta Cristina, Parla, Madrid
  - Hospital Madrid Norte Sanchinarro Centro Integral Oncológico Clara Campal Ensayos Clínicos, PAU de Sanchinarro, Madrid
  - Hospital Costa del Sol, Marbella, Malaga
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Centro Oncologico MD Anderson, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Switzerland (3):
  - Tumor Center Hirslanden Medical Center, Aarau
  - Spital STS AG Onkologiezentrum Thun - Berner Oberland, Thun
  - Kantonsspital Winterthur Medizinische Onkologie, Winterthur
- Chang Gung Medical Foundation, Linkou Branch, Taoyuan District, Taiwan
- Affinity Research Limited, Nassau, CB, The Bahamas
- Ege Universitesi Tip Fakultesi Tulay Aktas Onkoloji Hastanesi, Bornova, İzmir, Turkey (Türkiye)
- Ukraine (10):
  - Komunalnyy Zaklad Cherkasskyy Oblasnyy Onkologichnyy Dyspanser, Cherkassy
  - Chernivtsi Regional Oncology Centre Outpatient Department Bukovynian State Medical University Department of Oncology and Radiology, Chernivtsi
  - City Multifield Clinical Hospital, Dnipropetrovsk
  - Donetsk Regional Antitumor Center Department of Pretumor Diseases and Tumor Treatment, Donetsk
  - S.P. Grigoreva Institute of Medical Radiology Department of Chemotherapy, Kharkiv
  - National Institute of Cancer Department of Conseravtive Methods of Treatment, Kyiv
  - Volyn Regional Oncological Center, Lutsk
  - State Oncological Regional Treatment and Diagnostic Center, Lviv
  - Mariupil Oncological Center, Mariupil
  - Sumy Regional Clinical Oncology Centre, Sumy
- United Kingdom (2):
  - Guy's and St Thomas NHS Foundation Trust Management Offices 4th Floor Bermondsey Wing Guy's Hospital, London
  - Nottingham University Hospital, Nottingham

REFERENCES:
- [Derived] Awada A, Colomer R, Inoue K, Bondarenko I, Badwe RA, Demetriou G, Lee SC, Mehta AO, Kim SB, Bachelot T, Goswami C, Deo S, Bose R, Wong A, Xu F, Yao B, Bryce R, Carey LA. Neratinib Plus Paclitaxel vs Trastuzumab Plus Paclitaxel in Previously Untreated Metastatic ERBB2-Positive Breast Cancer: The NEfERT-T Randomized Clinical Trial. JAMA Oncol. 2016 Dec 1;2(12):1557-1564. doi: 10.1001/jamaoncol.2016.0237. PMID 27078022

RESULTS

PARTICIPANT FLOW:
Groups:
- Neratinib + Paclitaxel: Neratinib + Paclitaxel
  Neratinib: Neratinib - 240 mg orally daily, administered once daily. Treatment will be administered until documented disease progression, symptomatic deterioration, unacceptable toxicity, death or withdrawal of consent.
  Paclitaxel: Paclitaxel - 80 mg/m2 IV administered on days 1, 8, and 15 of a 28-day cycle. Treatment will be administered until documented disease progression, symptomatic deterioration, unacceptable toxicity, death or withdrawal of consent.
- Trastuzumab + Paclitaxel: Trastuzumab + Paclitaxel
  Trastuzumab: Trastuzumab - 4 mg/kg IV initial loading dose followed by subsequent once weekly doses of 2 mg/kg IV. Treatment will be administered until documented disease progression, symptomatic deterioration, unacceptable toxicity, death or withdrawal of consent.
  Paclitaxel: Paclitaxel - 80 mg/m2 IV administered on days 1, 8, and 15 of a 28-day cycle. Treatment will be administered until documented disease progression, symptomatic deterioration, unacceptable toxicity, death or withdrawal of consent.
Period: Overall Study
Arm/Group | Neratinib + Paclitaxel | Trastuzumab + Paclitaxel
Started | 242 | 237
Received Treatment | 240 | 234
Completed | 27 | 30
Not Completed | 215 | 207
Not completed — Death | 75 | 70
Not completed — Lost to Follow-up | 10 | 5
Not completed — Withdrawal by Subject | 38 | 27
Not completed — By Sponsor due to Protocol Amendment | 92 | 105

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neratinib + Paclitaxel | Trastuzumab + Paclitaxel | Total
Number analyzed (Participants) | 242 | 237 | 479
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 199 | 193 | 392
  >=65 years | 43 | 44 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (11.6) | 54.3 (11.0) | 54.1 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 242 | 237 | 479
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: Defined as the interval from the date of randomization until the first date on which recurrence or progression, or death due to any cause, is documented, censored at the last assessable evaluation or at the initiation of new anticancer therapy.
Time Frame: From randomization to disease progression or death, assessed up to 5.3 years
Population: all randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Neratinib + Paclitaxel | Trastuzumab + Paclitaxel
Number analyzed (Participants) | 242 | 237
months | 12.9 [11.1 to 14.9] | 12.9 [11.1 to 14.8]
Statistical Analysis 1: Comparison: Neratinib + Paclitaxel vs Trastuzumab + Paclitaxel; Test type: Superiority; p = 0.8934, Log Rank; Hazard Ratio (HR) = 1.015, 95% CI 2-sided [0.813 to 1.269]

2. Secondary Outcome: Objective Response Rate
Description: Defined as the percentage of subjects who achieved confirmed tumor response (complete or partial response) per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.0: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; and Non-Progressive Disease for non-target lesions, and no new lesions.
Time Frame: From randomization to disease progression or last tumor assessment, assessed up to 5.3 years
Population: all randomized patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neratinib + Paclitaxel | Trastuzumab + Paclitaxel
Number analyzed (Participants) | 242 | 237
percentage of participants | 74.8 [68.8 to 80.1] | 77.6 [71.8 to 82.8]
Statistical Analysis 1: Comparison: Neratinib + Paclitaxel vs Trastuzumab + Paclitaxel; Test type: Other; p = 0.5219, Mantel Haenszel; Risk Difference (RD) = 0.028, 95% CI 2-sided [-0.048 to 0.105]

3. Secondary Outcome: Duration of Response
Description: Measured from the time at which measurement criteria were first met for CR or PR (whichever status was recorded first), until the date of first recurrence, disease progression (PD), or death was objectively documented, taking as a reference for PD the smallest measurements recorded since enrollment, per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.0: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; and Non-PD for non-target lesions, and no new lesions.
Time Frame: From first response to first PD or death, assessed up to 5.3 years after first subject randomized
Population: patients who responded
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Neratinib + Paclitaxel | Trastuzumab + Paclitaxel
Number analyzed (Participants) | 181 | 184
months | 13.1 [11.1 to 15.4] | 12.9 [11.0 to 15.1]
Statistical Analysis 1: Comparison: Neratinib + Paclitaxel vs Trastuzumab + Paclitaxel; Test type: Other; p = 0.8431, Log Rank; Hazard Ratio (HR) = 0.974, 95% CI 2-sided [0.752 to 1.262]

4. Secondary Outcome: Clinical Benefit Rate
Description: Defined as the proportion of patients who achieved overall tumor response (CR or PR) or SD for at least 24 weeks per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.0: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; and Non-PD for non-target lesions, and no new lesions; Stable Disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: From randomization to disease progression or death, assessed up to 5.3 years
Population: all randomized patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neratinib + Paclitaxel | Trastuzumab + Paclitaxel
Number analyzed (Participants) | 242 | 237
percentage of participants | 88.4 [83.7 to 92.2] | 85.2 [80.1 to 89.5]
Statistical Analysis 1: Comparison: Neratinib + Paclitaxel vs Trastuzumab + Paclitaxel; Test type: Other; p = 0.2360, Mantel Haenszel; Risk Difference (RD) = -0.032, 95% CI 2-sided [-0.093 to 0.029]

5. Secondary Outcome: Symptomatic or Progressive Central Nervous System (CNS) Lesions
Description: Defined as the time interval from the date of randomization until the first date of CNS symptoms, the imaging examination shows CNS progression or is censored at the last assessable evaluation on study or prior to new anti-cancer therapy, if applicable.
  If median time to Symptomatic or Progressive CNS Lesions is not estimable, cumulative incidence will be reported instead.
Time Frame: From randomization to disease progression PD or last tumor assessment, assessed up to 5.3 years
Population: all randomized patients
Measure: Count of Participants; unit: Participants
Arm/Group | Neratinib + Paclitaxel | Trastuzumab + Paclitaxel
Number analyzed (Participants) | 242 | 237
Participants | 20 | 41
Statistical Analysis 1: Comparison: Neratinib + Paclitaxel vs Trastuzumab + Paclitaxel; Test type: Other; p = 0.0036, Log Rank; Hazard Ratio (HR) = 0.449, 95% CI 2-sided [0.259 to 0.780]

ADVERSE EVENTS:
Time Frame: From First Dose through 28 days after last dose, assessed up to 5.3 years
Groups:
- Neratinib+Paclitaxel: Neratinib + Paclitaxel
- Trastuzumab+Paclitaxel: Trastuzumab + Paclitaxel
Arm/Group | Neratinib+Paclitaxel | Trastuzumab+Paclitaxel
Serious Adverse Events (participants affected / at risk) | 67/240 | 56/234
Other Adverse Events (participants affected / at risk) | 239/240 | 230/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neratinib+Paclitaxel (N=240) | Trastuzumab+Paclitaxel (N=234)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Retinal degeneration (Eye disorders) | 1 | 0
Uveitis (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 2 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 12 | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 7 | 1
Adhesion (General disorders) | 1 | 0
Disease progression (General disorders) | 3 | 0
Fatigue (General disorders) | 1 | 1
Generalised oedema (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 1
Pyrexia (General disorders) | 3 | 5
Sudden death (General disorders) | 0 | 1
Swelling (General disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 2 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Contrast media allergy (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 1
Food allergy (Immune system disorders) | 1 | 0
Type IV hypersensitivity reaction (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Candida infection (Infections and infestations) | 1 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 6
Dengue fever (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 2 | 2
Empyema (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 3 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pleural infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 3
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Drug administration error (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
General physical condition abnormal (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 7 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 0
Cerebellar ischaemia (Nervous system disorders) | 0 | 1
Coma (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 4 | 0
Depression (Psychiatric disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 1
Prerenal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neratinib+Paclitaxel (N=240) | Trastuzumab+Paclitaxel (N=234)
Anaemia (Blood and lymphatic system disorders) | 75 | 65
Leukopenia (Blood and lymphatic system disorders) | 72 | 74
Lymphopenia (Blood and lymphatic system disorders) | 32 | 30
Neutropenia (Blood and lymphatic system disorders) | 77 | 79
Abdominal distension (Gastrointestinal disorders) | 16 | 4
Abdominal pain (Gastrointestinal disorders) | 51 | 26
Abdominal pain upper (Gastrointestinal disorders) | 30 | 18
Constipation (Gastrointestinal disorders) | 35 | 44
Diarrhoea (Gastrointestinal disorders) | 222 | 78
Dyspepsia (Gastrointestinal disorders) | 31 | 20
Haemorrhoids (Gastrointestinal disorders) | 4 | 12
Nausea (Gastrointestinal disorders) | 107 | 70
Stomatitis (Gastrointestinal disorders) | 59 | 46
Vomiting (Gastrointestinal disorders) | 87 | 37
Asthenia (General disorders) | 53 | 36
Fatigue (General disorders) | 77 | 64
Influenza like illness (General disorders) | 10 | 14
Oedema (General disorders) | 11 | 15
Oedema peripheral (General disorders) | 34 | 40
Pain (General disorders) | 13 | 13
Pyrexia (General disorders) | 41 | 44
Cystitis (Infections and infestations) | 13 | 12
Influenza (Infections and infestations) | 11 | 13
Nasopharyngitis (Infections and infestations) | 29 | 33
Paronychia (Infections and infestations) | 16 | 9
Rhinitis (Infections and infestations) | 2 | 12
Upper respiratory tract infection (Infections and infestations) | 26 | 32
Urinary tract infection (Infections and infestations) | 17 | 15
Alanine aminotransferase increased (Investigations) | 31 | 26
Aspartate aminotransferase increased (Investigations) | 26 | 22
Blood alkaline phosphatase increased (Investigations) | 15 | 11
Weight decreased (Investigations) | 38 | 12
Weight increased (Investigations) | 8 | 14
Decreased appetite (Metabolism and nutrition disorders) | 76 | 41
Dehydration (Metabolism and nutrition disorders) | 18 | 3
Hypercreatininaemia (Metabolism and nutrition disorders) | 13 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 16
Hypocalcaemia (Metabolism and nutrition disorders) | 19 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 23 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 | 44
Back pain (Musculoskeletal and connective tissue disorders) | 37 | 27
Bone pain (Musculoskeletal and connective tissue disorders) | 11 | 12
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17 | 12
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 13 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13 | 18
Myalgia (Musculoskeletal and connective tissue disorders) | 31 | 32
Pain in extremity (Musculoskeletal and connective tissue disorders) | 30 | 25
Dizziness (Nervous system disorders) | 52 | 30
Dysgeusia (Nervous system disorders) | 35 | 16
Headache (Nervous system disorders) | 49 | 45
Hypoaesthesia (Nervous system disorders) | 18 | 25
Neuropathy peripheral (Nervous system disorders) | 61 | 60
Paraesthesia (Nervous system disorders) | 21 | 12
Peripheral sensory neuropathy (Nervous system disorders) | 47 | 53
Insomnia (Psychiatric disorders) | 32 | 28
Breast pain (Reproductive system and breast disorders) | 5 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 47
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 28 | 22
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 36 | 20
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 18 | 20
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 17
Alopecia (Skin and subcutaneous tissue disorders) | 126 | 133
Dry skin (Skin and subcutaneous tissue disorders) | 14 | 12
Erythema (Skin and subcutaneous tissue disorders) | 9 | 16
Nail disorder (Skin and subcutaneous tissue disorders) | 33 | 31
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 14 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 19 | 22
Rash (Skin and subcutaneous tissue disorders) | 72 | 51
Hot flush (Vascular disorders) | 13 | 8
Hypertension (Vascular disorders) | 13 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less